CLINICAL TRIAL: NCT06941961
Title: Efficacy and Safety of Intermittent Theta Burst Stimulation in Acute Anterior Circulation Ischemic Stroke Patients Undergoing Mechanical Thrombectomy
Brief Title: iTBS for Acute Ischemic Stroke After Thrombectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iTBS-ACT
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS (Active Comparator): Patients are treated with intermittent theta burst stimulation (iTBS).
  Interventions: Device: intermittent theta burst stimulation
- sham-iTBS (Sham Comparator): Patients are treated with sham intermittent theta burst stimulation (sham-iTBS).
  Interventions: Device: sham intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — The iTBS delivered to the ipsilesional primary motor cortex (M1) at 80% resting motor threshold (RMT). Each session consists of 600 pulses (3-minute trains of 50 Hz triplets repeated every 10 seconds, twice daily with a 5-minute interval), administered for 7 consecutive days starting within 6 hours post-randomization.
  Arms: iTBS
Device: sham intermittent theta burst stimulation — Sham-iTBS is performed in the same way as the treatment group but uses 20% RMT.
  Arms: sham-iTBS

SUMMARY:
The goal of this randomized, single-blind, parallel-controlled clinical trial is to evaluate the efficacy and safety of intermittent theta burst stimulation (iTBS) as an adjunctive therapy for acute anterior circulation ischemic stroke patients who have undergone successful mechanical thrombectomy (MT). The study population includes adults aged 18-85 with NIHSS scores 5-25 post-MT and eTICI≥2b reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-85 years, regardless of gender.
* 2) Acute ischemic stroke caused by occlusion of the anterior circulation large vessels (internal carotid artery, M1 or M2 segment of the middle cerebral artery), verified by CTA or DSA.
* 3) Mechanical thrombectomy (MT) performed within 24 hours of symptom onset.
* 4) Successful Reperfusion: Post-MT eTICI score ≥ 2b.
* 5) NIHSS score 5-25 at 24 hours post-MT, with ≥2 points in at least one limb.

Exclusion Criteria:

* 1) Pre-stroke modified Rankin Scale (mRS) score ≥2.
* 2) PH2-type intracranial hemorrhage on brain CT post-MT.
* 3) Patients who underwent intracranial stent placement during MT.
* 4) Contraindications to iTBS: History of epilepsy or seizures, implanted cardiac pacemakers, cochlear implants, or other electronic/magnetic-sensitive devices.
* 5) Severe consciousness impairment, cognitive dysfunction, or psychiatric disorders preventing compliance with iTBS.
* 6) Expected survival <3 months due to other medical conditions or inability to complete follow-up for any reason.
* 7) Participation in another interventional study.
* 8) Any other condition deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 at 90 days | 90 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
Distribution of Modified Rankin Scale (mRS) Scores at 90 Days | 90 days
  mRS scores (0-6) assess functional independence, where lower scores indicate better outcomes.
Distribution of Modified Rankin Scale (mRS) Scores at 30 Days | 30 days
  mRS scores (0-6) assess functional independence, where lower scores indicate better outcomes.
Differences in National Institutes of Health Stroke Scale (NIHSS) Score at 7 days | 7 days
  NIHSS (0-42) measures neurological deficit severity, with lower scores indicating better function.
Proportion of Patients with Early Neurological Deterioration (END) Within 7 Days | 7 days
  END is defined as an increase in NIHSS score ≥4 points from baseline.
All-Cause Mortality Rate at 90 Days | From randomization to 90 days
  Proportion of patients who died from any cause within 90 days.
Incidence of Intracranial Hemorrhage (ICH) and Symptomatic ICH (sICH) During Intervention | 7 days
  ICH is assessed via imaging
Rate of iTBS-Related Adverse Events | From randomization to 90 days
  Includes seizures, headache, scalp discomfort, or other stimulation-related AEs.
Overall Adverse Event (AE) Rate | From randomization to 90 days
  Proportion of patients experiencing any AE during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China